CLINICAL TRIAL: NCT02542709
Title: The Use of Noninvasive Brain Stimulation in Post-traumatic Stress Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2013-011; 2013-341 (Other: Institut de réadaptation en déficience physique de Québec)
Record Dates: First submitted 2015-03-26; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active transcranial magnetic stimulation (Active Comparator): Active transcranial magnetic stimulation will induce real pulses using the transcranial magnetic stimulation device.
  Interventions: Device: Active repetitive Transcranial Magnetic Stimulation
- Sham transcranial magnetic stimulation (Sham Comparator): Sham transcranial magnetic stimulation will not induce any pulses using the same transcranial magnetic stimulation device but by also adding a sham block device.
  Interventions: Device: Sham repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Active repetitive Transcranial Magnetic Stimulation — Active transcranial magnetic stimulation will induce real pulses using the transcranial magnetic stimulation device.
  Arms: Active transcranial magnetic stimulation
Device: Sham repetitive Transcranial Magnetic Stimulation — Sham transcranial magnetic stimulation will not induce any pulses using the same transcranial magnetic stimulation device but by also adding a sham block device.
  Arms: Sham transcranial magnetic stimulation

SUMMARY:
The purpose of this trial is to study the effect of noninvasive brain stimulation in adults with post-traumatic stress disorder.

DETAILED DESCRIPTION:
The purpose of this trial is to study the effect of noninvasive brain stimulation on symptoms severity in adults with post-traumatic stress disorder.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old

Exclusion Criteria:

* Transcranial magnetic stimulation ineligibility

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Severity of symptoms on the following clinical scale: PTSD symptoms as assessed by the Modified PTSD Symptom Scale (MPSS-SR) | 2 months
  Units will be the differences (%) in scores before and after the intervention

SECONDARY OUTCOMES:
Severity of symptoms on the following clinical scale: anxiety symptoms as assessed by the Beck Anxiety Inventory (BAI) | 2 months
  Units will be the differences (%) in scores before and after the intervention
Severity of symptoms on the following clinical scale: depression symptoms as assessed by the Beck Depression Inventory (BDI) | 2 months
  Units will be the differences (%) in scores before and after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- IRDPQ, Québec, Canada